CLINICAL TRIAL: NCT01996033
Title: This is a Post Market, Multi-center, Open Label, Observational Study. Approximately 500 Subjects With Uncontrolled Hypertension Will Undergo Renal Artery Ablation
Brief Title: EnligHTN German Observational Study of Renal Denervation for Uncontrolled Hypertension
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CV-12-064-GE-HT
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Uncontrolled Hypertension
Keywords: uncontrolled hypertension; Renal Denervation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to further evaluate the safety and performance of the EnligHTN™ Renal Denervation System in the treatment of patients with uncontrolled hypertension in clinical routine practice.

DETAILED DESCRIPTION:
This is a post market, multi-center, open label, observational study. Approximately 500 subjects with uncontrolled hypertension will undergo renal artery ablation at approximately 40 investigational sites located in Germany and will be followed for 1 year post procedure.The expected duration of the investigation will be approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject is planned to undergo a renal denervation procedure for the treatment of hypertension
* Subject is ≥18 years of age at time of consent
* Subject must be able and willing to provide written informed consent
* Subject must be able and willing to comply with the required follow-up schedule
* Subject has office Systolic Blood Pressure (SBP) ≥ 140 mmHg
* Subject has established hypertension (diagnosed ≥12 months prior to baseline) and is on a guideline based drug regimen at a stable (≥ 14 days) and a fully tolerated dose consisting of ≥3 anti-hypertensive medications (including 1 diuretic), or subject has documented drug intolerance to 2 or more of the 4 major classes of anti-hypertensives (ACE-I/ Angiotensin Receptor Blocker (ARB), Calcium Channel Blockers, Beta Blockers, or diuretic) and is unable to take 3 anti-hypertensive drugs

Exclusion Criteria:

* Subject has known significant renovascular abnormalities such as renal artery stenosis > 30%
* Subject has undergone prior renal angioplasty, renal denervation, indwelling renal stents, and/or abdominal aortic stent grafts
* Subject has a history of hemodynamically significant valvular heart disease
* Subject has blood clotting abnormalities
* Subject life expectancy is < 12 months, as determined by the Study Investigator
* Subject is participating in another clinical study which has the potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population enrolled in this investigation will consist of males and females with uncontrolled hypertension who meet all inclusion criteria, and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph K Naber, MD, Principal Investigator — Elisabeth-Krankenhaus Essen, Germany
Locations (12):
- Germany (12):
  - Kliniken Villingen-Schwenningen, Villingen-Schwenningen, Baden-Wurttemberg
  - Kliniken Oberallgäu gGmbH Klinik Immenstadt, Immenstadt im Allgäu, Bavaria
  - Immanuelklinikum Bernau und Herzzentrum Brandenburg, Bernau bei Berlin, Brandenburg
  - Klinikum Ernst von Bergmann, Potsdam, Brandenburg
  - Asklepios Schwalm-Eder-Kliniken GmbH, Schwalmstadt, Hesse
  - Klinikum Oldenburg gGmbH, Oldenburg, Lower Saxony
  - Medizinische Einrichtungen der Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Elisabeth-Krankenhaus Essen, Essen, North Rhine-Westphalia
  - Kardiologische Praxis Wuppertal, Wuppertal, North Rhine-Westphalia
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Augusta-Krankenhaus Düsseldorf, Düsseldorf
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Schwäbisch Hall

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Full Cohort: All subjects - this is a single arm study
Period: Overall Study
Arm/Group | Full Cohort
Started | 25
Completed | 16
Not Completed | 9
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: All subjects
Arm/Group | Full Cohort
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Years since HTN diagnosis [Mean (Standard Deviation); unit: years] — Population: Some subjects were missing baseline data.
  years
    number analyzed (Participants) | 17
    (all) | 19.2 (15.5)
Years taking anti-HTN medications [Mean (Standard Deviation); unit: years] — Population: Some subjects were missing baseline data.
  years
    number analyzed (Participants) | 12
    (all) | 15.4 (11.3)
Myocardial Infarction [Count of Participants; unit: Participants] | 2
Coronary Artery Disease [Count of Participants; unit: Participants] | 7
Coronary Artery Bypass Graft [Count of Participants; unit: Participants] | 3
Percutaneous Coronary Intervention [Count of Participants; unit: Participants] | 2
Cerebrovascular Accident [Count of Participants; unit: Participants] | 3
Obstructive Sleep Apnea [Count of Participants; unit: Participants] | 7
Diabetes (Type II) [Count of Participants; unit: Participants] | 13
Smoker [Count of Participants; unit: Participants] | 8
Weight [Mean (Standard Deviation); unit: kilograms] | 88.0 (18.7)
Height [Mean (Standard Deviation); unit: centimeters] | 171.2 (8.4)
BMI [Mean (Standard Deviation); unit: kilograms/meter2] | 29.9 (5.6)
Office Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 164.5 (20.2)
  Diastolic | 87.8 (12.6)
24Hr Ambulatory Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Some subjects were missing baseline data.
  mmHg
    Systolic: number analyzed (Participants) | 18
    Systolic | 157.1 (18.6)
    Diastolic: number analyzed (Participants) | 18
    Diastolic | 83.2 (15.7)
Serum Creatinine [Mean (Standard Deviation); unit: micromoles/liter] | 88.6 (18.7)
Estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: mL/min per 1.73m2] | 72.8 (16.1)
Number of Antihypertensive Medications [Mean (Standard Deviation); unit: medications] | 4.7 (1.1)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Population: Some subjects were missing baseline data.
  beats per minute
    number analyzed (Participants) | 22
    (all) | 71.2 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction in Office Systolic Blood Pressure at 6 Months
Description: Positive number indicates a reduction (improvement) in blood pressure
Time Frame: 6 months
Population: All subjects with data available at baseline and 6-month follow up
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Full Cohort
Number analyzed (Participants) | 15
mmHg | 17.6 (21.5)

2. Other Pre Specified Outcome: Reduction in Office Diastolic Blood Pressure
Description: Positive number indicates a reduction (improvement) in blood pressure
Time Frame: 6 Months
Population: Subjects with baseline and follow up data available
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Full Cohort
Number analyzed (Participants) | 15
mmHg | 9.9 (11.9)

3. Other Pre Specified Outcome: Reduction in Office Diastolic Blood Pressure
Description: Positive number indicates a reduction (improvement) in blood pressure
Time Frame: 12 Months
Population: Subjects with baseline and follow up data available
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Full Cohort
Number analyzed (Participants) | 14
mmHg | 3.6 (17.3)

4. Other Pre Specified Outcome: Reduction in Office Systolic Blood Pressure
Description: Positive number indicates a reduction (improvement) in blood pressure
Time Frame: 12 Months
Population: Subjects with baseline and follow up data available
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Full Cohort
Number analyzed (Participants) | 14
mmHg | 7.0 (26.0)

5. Other Pre Specified Outcome: Reduction in 24 Hour Ambulatory Systolic Blood Pressure
Description: Positive number indicates a reduction (improvement) in blood pressure
Time Frame: 12 Months
Population: Subjects with baseline and follow up data available
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Full Cohort
Number analyzed (Participants) | 12
mmHg | 14.6 (13.7)

6. Other Pre Specified Outcome: Reduction in 24 Hour Ambulatory Diastolic Blood Pressure
Description: Positive number indicates a reduction (improvement) in blood pressure
Time Frame: 12 Months
Population: Subjects with baseline and follow up data available
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Full Cohort
Number analyzed (Participants) | 12
mmHg | 6.7 (10.1)

7. Other Pre Specified Outcome: Proportion of Subjects Achieving <140mmHg Office Systolic Blood Pressure
Description: Positive number indicates a reduction (improvement) in blood pressure
Time Frame: 1 Month
Population: Subjects with baseline and follow up data available
Measure: Count of Participants; unit: Participants
Arm/Group | Full Cohort
Number analyzed (Participants) | 20
Participants | 8

8. Other Pre Specified Outcome: Proportion of Subjects Achieving <140mmHg Office Systolic Blood Pressure
Description: Positive number indicates a reduction (improvement) in blood pressure
Time Frame: 6 Months
Population: Subjects with baseline and follow up data available
Measure: Count of Participants; unit: Participants
Arm/Group | Full Cohort
Number analyzed (Participants) | 15
Participants | 6

9. Other Pre Specified Outcome: Proportion of Subjects Achieving <140mmHg Office Systolic Blood Pressure
Description: Positive number indicates a reduction (improvement) in blood pressure
Time Frame: 12 Months
Population: Subjects with baseline and follow up data available
Measure: Count of Participants; unit: Participants
Arm/Group | Full Cohort
Number analyzed (Participants) | 14
Participants | 3

10. Other Pre Specified Outcome: Change in Estimated Glomerular Filtration Rate (eGFR)
Description: Change from baseline in eGFR
Time Frame: 12 Months
Population: Subjects with both baseline and follow up data available
Measure: Mean (Standard Deviation); unit: mL/min per 1.73m2
Arm/Group | Full Cohort
Number analyzed (Participants) | 9
mL/min per 1.73m2 | 3.8 (10.8)

ADVERSE EVENTS:
Arm/Group | Full Cohort
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Cohort (N=25)
Prostate Disease (Reproductive system and breast disorders) | 1 (1)
Arterial Hypertension/Hypertension (Vascular disorders) | 1 (2)
Multiple Organ Failure (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 1 (1)
VASC Vessel Stenosis (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Cohort (N=25)
Arterial Hypertension/Hypertension (Vascular disorders) | 2 (2)
Abnormal Lab Value (Suspicion of Cholangitis) (Hepatobiliary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Artery Stenosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less